CLINICAL TRIAL: NCT06701669
Title: Phase 2 Clinical Platform Trial Investigating Multiple Therapeutic Options for the Treatment of Hospitalized Patients With Acute Respiratory Distress Syndrome (ARDS)
Brief Title: JUST BREATHE, Breathing Life Into Innovative Therapies for ARDS- Cohort B: Paridiprubart
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: PPD Development, LP (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency); InflaRx GmbH (Industry); Edesa Biotech Inc. (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BP-ARDS-P2-001 (paridiprubart); 75A50124C00001 (Other Grant/Funding Number: Biomedical Advanced Research and Development Authority (BARDA))
Record Dates: First submitted 2024-11-20; First posted 2024-11-22 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Acute Respiratory Distress Syndrome (ARDS); ARDS; ARDS (Acute Respiratory Distress Syndrome); Acute Respiratory Distress Syndrome
Keywords: BARDA; JUST BREATHE; ARDS; Acute Respiratory Distress Syndrome; Acute Respiratory Failure
MeSH Terms: conditions — Respiratory Distress Syndrome; Acute Lung Injury

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: The overall 2-step randomization scheme will be implemented.
  * Randomization Level 1 will be open-label, assigning an eligible patient to one of the available treatment cohorts.
  * Randomization Level 2 will be double-blinded and will randomize participants at a 1:1 ratio to receive either IP or placebo within a specific cohort. Thus, the PPD blinded team, site blinded staff members, and participants/legal authorized representative will be considered blinded to study treatment assignment (either IP or placebo) throughout the course of the study.
  To preserve the integrity of the study blind, an unblinded pharmacist at each site will be responsible for the reconstitution and dispensation of all study drugs and placebos and will endeavor to ensure that there are no observable differences between the treatment groups (IP or placebo) when dispensing the study materials.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort B: paridiprubart (Experimental)
  Interventions: Drug: Cohort B: paridiprubart
- Cohort B: placebo (Placebo Comparator)
  Interventions: Drug: Cohort B: placebo

INTERVENTIONS:
Drug: Cohort B: paridiprubart — Administered as a single IV dose of 15 mg/kg up to maximum of 1440 mg on Day 1
  Arms: Cohort B: paridiprubart
Drug: Cohort B: placebo — Administered as a single IV dose of placebo on Day 1
  Arms: Cohort B: placebo

SUMMARY:
This is a Phase 2 multicenter, randomized, double-blinded, placebo-controlled study that will evaluate the safety and efficacy of host-directed therapeutics in hospitalized adults diagnosed with Acute Respiratory Distress Syndrome (ARDS) utilizing a platform trial design.

Cohort B: Participants will be randomized to receive either a placebo or paridiprubart.

This record describes the default procedures and analyses for Cohort B. Please see NCT06703073 for information on the BP-ARDS-P2-001 Master Protocol.

DETAILED DESCRIPTION:
This is a master protocol for a Phase 2 platform clinical trial to evaluate host-directed therapeutic candidates (i.e., investigational product, IP) for the treatment of hospitalized participants diagnosed with ARDS. The safety and efficacy of each IP will be studied within its own cohort (IP versus Placebo). All patients will continue to receive standard treatments for ARDS as per the investigator. An individual participant will complete the study in approximately 90 days. The study will include a screening period (<24 hours from providing informed consent to treatment), in-hospital treatment period with IP/placebo starting on Day 1 through discharge from the hospital, and a follow-up period after discharge from the hospital through the end of study (Day 90 + 2 weeks). Outcome data will be assembled for each patient over time (such as ventilatory status, oxygenation, and survival). Functional status using the WHO Ordinal scale and Karnofsky scale will be collected. Resource utilization will be calculated (length of stay in a critical care setting, days intubated, and survival).

All participants will undergo a series of physical exams, laboratory assessments/biomarker collections, ECG, Chest X-ray or CT scan, and questionnaires through Day 90. Exploratory biomarkers will be evaluated over time to facilitate clinical learning. This record only includes information relevant to the paridiprubart cohort.

ELIGIBILITY:
Inclusion Criteria:

The following inclusion criteria are in addition to the exclusion criteria specified in the Master Protocol NCT06703073:

- ARDS Severity of moderate or severe based on PaO2/FiO2 or SpO2/FiO2 assessment at the time of randomization.

Exclusion Criteria:

The following exclusion criteria are in addition to the exclusion criteria specified in the Master Protocol NCT06703073.

-Participant has a known allergy or known hypersensitivity to paridiprubart or its excipients, including polysorbate 80

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-06-10 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality (ACM) rate at Day 28 | Day 28

SECONDARY OUTCOMES:
ACM at Day 60 and Day 90 | Day 60 and Day 90
ACM+ at Day 28, Day 60, and Day 90 | Day 28, Day 60, and Day 90
  ACM+ composite score will be constructed by combining ACM and participant-relevant, infection-related Adverse Events (AE) from the MedDRA toxic/septic shock standardized MedDRA queries.
Improvements in oxygenation measured as change from baseline in PaO2/FiO2 ratio up to and including Day 28 (or discharge, whichever is earlier) | Up to and including Day 28 or until Discharge (whichever is earlier)
Incidence of new invasive mechanical ventilation use during the study up to and including Day 28 | Up to and including Day 28
Ventilator-free days up to and including Day 28 | Up to and including Day 28
Proportion of participants alive and free of mechanical ventilation at Days 28, 60, and 90 | Days 28, 60, and 90
Time to recover gas exchange to a PaO2/FiO2 ≥ 300 measured on 2 consecutive days during the first 28 days after informed consent | Up to and including Day 28
Extracorporeal Membrane Oxygenation (ECMO) free days up to and including Day 28 | up to and including Day 28
Incidence of participants with new ECMO use during the study up to and including Day 28 | up to and including Day 28
Proportion of participants alive and free of ECMO at Days 28, 60, and 90 | Days 28, 60, and 90
Proportion of participants achieving a ≥2-point improvement from baseline in the World Health Organization (WHO) 8-levels ordinal scale (from 0-8) | While Hospitalized (up to 90 days)
Time to an improvement of one category and two categories from baseline using the WHO 8-levels ordinal scale (from 0-8) at Days 28, 60, and 90 (while hospitalized) | While Hospitalized (up to 90 days)
Mean change in the WHO 8-levels ordinal scale from baseline through Day 90 (while hospitalized) | While Hospitalized (up to 90 days)
Proportion of participants who improve clinical status as measured by the Karnofsky scale | Post hospitalization through Day 90
  The Karnofsky scale is used to assess the general condition of the patient. Scores range from 0 to 100 with higher scores indicating better functional ability.
Days of hospitalization up to and including Day 28 | up to and including Day 28
Days of ICU stay up to and including Day 28 | up to and including Day 28
Change in Short Form Health Survey (SF-12) from hospital discharge to Day 60 and to Day 90 | from hospital discharge to Day 60 and to Day 90
  The SF-12 is a self-reported outcome measure composed by 12 items which examine eight dimensions of physical and mental health. Scores range from 0 to 100, with higher scores indicating better physical and mental health functioning.
Change in St. George's Respiratory Questionnaire (SGRQ) from hospital discharge to Day 60 and to Day 90 | From hospital discharge to Day 60 and to Day 90
  The SGRQ comprises of 50 items and consists of two parts. The first part pertains to symptoms and the second pertains to functional status as well as social and psychological impact of disease. Overall scores range between 0 and 100 with higher scores indicating more limitations.
Incidence and severity of adverse events (AEs) /adverse event of special interest (AESI) / serious adverse event (SAEs) | Through Day 90

CONTACTS AND LOCATIONS:
Locations (30):
- United States (30):
  - Community Regional Medical Center, Fresno, California
  - Long Beach Memorial Medical Center, Long Beach, California
  - University of California Irvine Medical Center, Orange, California
  - University of California Davis Medical Center - Pulmonary Medicine, Sacramento, California
  - Denver Health Hospital and Authority, Denver, Colorado
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Nova Clinical Research, Bradenton, Florida
  - North Florida / South Georgia Veterans Health System, Gainesville, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - St. Luke's Boise Medical Center, Boise, Idaho
  - OSF Saint Francis Medical Center-, Peoria, Illinois
  - Tufts Medical Center, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - University of Michigan Hospital, Ann Arbor, Michigan
  - Henry Ford Health Hospital, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Renown Institute for Heart & Vascular Health, Reno, Nevada
  - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Montefiore Hospital - Moses Campus, The Bronx, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Durham VA Medical Center, Durham, North Carolina
  - Mercy Health - St. Vincent Medical Center, Toledo, Ohio
  - The University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor All Saints Medical Center, Fort Worth, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Intermountain Medical Center, Murray, Utah
  - Swedish Medical Center, Seattle, Washington